CLINICAL TRIAL: NCT03203382
Title: Corneal Nerve Structure in Sjogren's
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 823009
Record Dates: First submitted 2017-01-04; First posted 2017-06-29 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Sjogren's Syndrome; Vitamin D Deficiency
MeSH Terms: conditions — Sjogren's Syndrome; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients who are suspected of or diagnosed with Sjogren's disease will be evaluated for ocular symptoms and corneal nerve morphology. We are specifically interested in the relationship between Vitamin D level and aberrations in the morphology of the corneal nerves.

DETAILED DESCRIPTION:
Patients with either suspected or confirmed diagnosis of Sjogren's disease will be recruited to participate. Participation will involve the completion of a brief survey (the OSDI), corneal evaluation with an aesthesiometer, corneal staining with fluorescein and lissamine green, and finally measurement of tear-film breakup time. In addition, participants will have their corneal nerve morphology evaluated with the Heidelberg confocal microscope and finally they will have a blood draw performed to assess vitamin D level.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed Sjogren's syndrome
* 18+ years of age

Exclusion Criteria:

* Any condition that in the opinion of the investigator may confound study results or cause concerns for safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected or confirmed Sjogren's patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Corneal Nerve Morphology | one time exam
  Heidelberg Retina Tomograph with the Rostock Cornea Module
Vitamin D Level | one time exam at baseline, day 1
  serum

SECONDARY OUTCOMES:
vital dye staining | one time exam at baseline, day 1
  corneal staining

CONTACTS AND LOCATIONS:
Overall Officials: Giacomina Massaro-Giordano, Principal Investigator — Scheie Eye Institute
Locations (1):
- Scheie Eye Institute of the University of Pennsylvania, Philadelphia, Pennsylvania, United States